CLINICAL TRIAL: NCT03254784
Title: A Phase 1, Randomized, Open-Label, Single-Dose, Crossover Study To Evaluate the Bioavailability of BMS-986165 Tablet Formulation Relative To BMS-986165 Capsule Formulation and the Effect of a High-Fat/ High-Calorie Meal And Increased Gastric pH on the Bioavailability of BMS-986165 Tablet Formulation in Healthy Subjects
Brief Title: A Study to Evaluate BMS-986165 Tablet Formulation Relative to BMS-986165 Capsule Formulation and the Effect of a High-Fat/ High-Calorie Meal and Increased Gastric pH on the BMS-986165 Tablet Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IM011-031
Record Dates: First submitted 2017-08-17; First posted 2017-08-18 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Systemic Lupus Erythematosus; Arthritic Psoriasis; Psoriasis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis, Psoriatic; Psoriasis; Inflammatory Bowel Diseases | interventions — deucravacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Tablet-Capsule Crossover 1 (Experimental): Variations between arms dependent on timing, fasting, dose and receiving the tablet or capsule at different treatment period combinations
  Interventions: Drug: BMS-986165 Capsule; Drug: BMS-986165 Tablet
- Tablet-Capsule Crossover 2 (Experimental): Variations between arms dependent on timing, fasting, dose and receiving the tablet or capsule at different treatment period combinations
  Interventions: Drug: BMS-986165 Capsule; Drug: BMS-986165 Tablet
- Tablet-Capsule Crossover 3 (Experimental): Variations between arms dependent on timing, fasting, dose and receiving the tablet or capsule at different treatment period combinations
  Interventions: Drug: BMS-986165 Capsule; Drug: BMS-986165 Tablet
- Tablet-Capsule Crossover 4 (Experimental): Variations between arms dependent on timing, fasting, dose and receiving the tablet or capsule at different treatment period combinations
  Interventions: Drug: BMS-986165 Capsule; Drug: BMS-986165 Tablet
- Tablet-Capsule Crossover 5 (Experimental): Variations between arms dependent on timing, fasting, dose and receiving the tablet or capsule at different treatment period combinations
  Interventions: Drug: BMS-986165 Capsule; Drug: BMS-986165 Tablet
- Tablet-Capsule Crossover 6 (Experimental): Variations between arms dependent on timing, fasting, dose and receiving the tablet or capsule at different treatment period combinations
  Interventions: Drug: BMS-986165 Capsule; Drug: BMS-986165 Tablet

INTERVENTIONS:
Drug: BMS-986165 Capsule — Oral capsule
Drug: BMS-986165 Tablet — Oral tablet

SUMMARY:
The purpose of this study is to evaluate BMS-986165 tablet formulation versus BMS-986165 capsule formulation. This study will also evaluate the effect of a high-fat/ high-calorie meal and increased gastric pH on the BMS-986165 tablet formulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be willing and able to complete all study-specific procedures and visits
* Healthy patients, as determined by no clinically significant deviation from normal in medical history, physical examination, electrocardiogram, and clinical laboratory determinations
* Body mass index (BMI) of 18 to 32 kg/m2, inclusive, at screening
* Normal renal function at screening

Exclusion Criteria:

* Women of childbearing potential not using an effective contraceptive method or are breastfeeding
* Any significant acute or chronic medical illness
* History of chronic headaches, defined as occurring 15 days or more a month, over the previous 3 months
* History of headaches related to caffeine withdrawal, including energy drinks
* History of syncope, orthostatic instability, or recurrent dizziness
* Active TB requiring treatment or documented latent TB within the previous 3 years

Other protocol defined inclusion/exclusion criteria could apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2017-11-04 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) derived from plasma concentration versus time | 5 days
AUC from time zero extrapolated to infinity [AUC(INF)] derived from plasma concentration versus time | 5 days
Area under the plasma concentration-time curve (AUC) from time zero to time of last quantifiable concentration [AUC(0-T)] derived from plasma concentration versus time | 5 days
Time of maximum observed plasma concentration (Tmax) derived from plasma concentration versus time | 5 days

SECONDARY OUTCOMES:
Adverse events measured by incidence | 26 days
Serious adverse events measured by incidence | Approximately 55 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PRA Health Sciences, Lenexa, Kansas, United States

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx